CLINICAL TRIAL: NCT06819137
Title: Evaluation of Gummy Smile With Artificial ıntelligence
Brief Title: Gummy Smile and Artificial Intelligence
Status: Active, not recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zeynep Turgut Çankaya, Gazi University, Gazi University
Other Study IDs: 13.02.2024/03
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Gummy Smile

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High gingival line: Gingival visibility exceeding 3 mm during smiling.
  Interventions: Other: Gingival visibility exceeding 3 mm during smiling

INTERVENTIONS:
Other: Gingival visibility exceeding 3 mm during smiling — Obtaining gummy smile photographs in accordance with the inclusion criteria specified in the study's materials and methods section.

SUMMARY:
A smile, as a nonverbal communication tool, is based on a balanced relationship between the teeth and the surrounding hard and soft tissues. The literature highlights the need for the evaluation of smile design using artificial intelligence (AI), suggesting that AI-assisted assessments could play a crucial role in all relevant stages of clinical parameters associated with gingival smile analysis. A gummy smile (GS) is defined as the excessive display of gingival tissue exceeding 3 mm during smiling.

The hypothesis of this study is based on the assumption that clinical data obtained for the analysis and diagnosis of gingival visibility can be accurately and reliably evaluated using AI-supported algorithms. To date, no study has been found in the literature that diagnoses GS using AI, predicts its etiological factors, and assesses its implications for treatment planning.

DETAILED DESCRIPTION:
Detailed Description

Among the causes of gummy smile (GS) are:

Excessive vertical development of the anterior maxilla Hyperactivity of the perioral muscles, leading to excessive lip elevation during smiling Short clinical crown length, which increases susceptibility to GS Altered passive eruption, gingival inflammation, and gingival hyperplasia contribute to a reduced clinical crown length. Cases where the vertical dimension of the teeth is shorter than the horizontal dimension suggest that passive eruption is a contributing factor to GS.

The extent of GS is not homogenous across all teeth involved in the smile and often results from multiple etiological factors. When gingival display is 3 mm, it is attributed solely to excessive gingival tissue. If an additional 2.2 mm of gingival display is present (3 mm + 2.2 mm), vertical maxillary excess (VME) is considered a contributing factor. When an additional 2.8 mm of gingival display is observed (3 mm + 2.2 mm + 2.8 mm), a hypermobile (HM) lip is implicated.

For instance:

A 3 mm GS over the maxillary left central incisor may be due to HM lip alone

A ≥8 mm GS over the maxillary left second premolar may result from a combination of:

HM lip (2.8 mm) Excessive gingival tissue (3 mm) VME (2.2 mm) This highlights the importance of measuring GS at each tooth level for accurate diagnosis and personalized treatment planning.

Assessing asymmetric GS requires individual measurements for each tooth, which can increase error likelihood and patient chair time. Given the significance of scientific research in identifying personalized intervention strategies for esthetic smile design, artificial intelligence (AI) could help transform the subjective nature of aesthetic perception into an individualized, scientific framework by adhering to specific reference parameters. The use of precise and valid measurements in GS evaluation can facilitate:

Diagnosis Etiological assessment Treatment planning By establishing a comprehensive dataset, the contributions of various etiologies can be analyzed by comparing measured variables with ideal reference values. A meticulous analysis of etiopathogenetic factors and the severity of the condition can be achieved through such an approach. Previous research indicates a need for more studies validating the accuracy and sensitivity of GS diagnosis and its etiological assessment.

AI-Based Analysis and Dataset Formation To date, no study has been found in the literature evaluating gingival display using AI. Unlike studies that use test datasets or publicly available open-access datasets for accuracy scoring, the data obtained in this research are exclusively derived from a training dataset.

To optimize the validation strategy of the AI model, selected clinical metrics were measured separately for each tooth involved in GS. Labeling was performed using a licensed web-based annotation platform that allows for multiple annotation options.

This study will include patients with a high smile line, selected from those who apply to the Department of Periodontology, Faculty of Dentistry, Gazi University. The labeling of patient photographs will be performed by two researchers:

A periodontologist A senior expert in artificial intelligence (AI) & software development Photographs of patients with gummy smile (GS) will be used to create training, validation, and test datasets.

Methodology for Dataset Formation

The simple random sampling method was used, with:

Confidence level: 0.95 Prevalence: 0.1 Margin of error: 0.05

The formation of these datasets will follow the steps outlined below:

A literature review was conducted to identify standardization methods for gingival visibility measurements. However, no standardized ruler system was found that allows for simultaneous calibration and measurement of gingival display across multiple teeth. Consequently, the need to develop a custom-designed ruler system specifically for this research emerged.

AI Model Training and Data Processing

Gingival display will be determined using a hybrid model. The training process will include:

Pixel Accuracy (PA) Mean Intersection over Union (mIoU) metrics

The dataset will be divided into:

Training set Validation set Testing set

Image preprocessing will include:

Resizing Normalization Transformation into tensors

ELIGIBILITY:
Inclusion Criteria:

Participants aged between 18 and 55 years.

Gingival Display During Smiling:

Presence of more than 3 mm of gingival display above the maxillary anterior teeth during smiling.

Gummy smile severity exceeding a predefined threshold, categorized as mild, moderate, or severe.

Oral and Periodontal Health:

Periodontally healthy individuals or those with minimal gingival inflammation. Anterior teeth free of caries or extensive restorations that may affect esthetic evaluation.

Participants with Class I occlusion or mild malocclusion.

Presence of etiological factors contributing to gummy smile, such as:

Vertical maxillary excess (VME) Hyperactive upper lip Altered passive eruption

History of Orthodontic or Surgical Treatment:

No history of previous gummy smile correction treatments. No orthodontic treatment or surgical intervention within the last 6-12 months.

Systemic Health and Medication Use:

Absence of systemic diseases or medication use that could influence gingival display.

Image Quality Requirements:

High-resolution and standardized photographs or video recordings. Images captured under consistent lighting conditions and fixed angles to ensure accurate evaluation of gingival display.

Exclusion Criteria:

Periodontal and Dental Conditions:

Presence of severe periodontal disease (e.g., periodontitis, gingival hyperplasia).

Extensive carious lesions, large restorations, or prosthetic crowns on anterior teeth.

History of traumatic dental injuries affecting the maxillary anterior region.

Occlusal and Skeletal Anomalies:

Severe malocclusion (e.g., Class II or III, open bite, crossbite). Jaw deformities requiring orthognathic surgery.

History of Previous Treatment for Gummy Smile:

Prior orthodontic treatment, periodontal surgery, or botulinum toxin injections for gummy smile correction.

History of orthognathic or maxillofacial surgery altering gingival display.

Systemic Health Conditions and Medication Use:

Presence of systemic diseases that could affect gingival tissue or facial muscle function (e.g., diabetes, neuromuscular disorders).

Use of medications known to induce gingival overgrowth, such as:

Calcium channel blockers Phenytoin Cyclosporine

Inadequate Image Quality for AI Analysis:

Low-resolution, blurred, or poorly standardized photographs. Inconsistent lighting conditions or improper facial positioning in images.

Pregnancy and Hormonal Influence:

Pregnant or postpartum individuals, as hormonal changes may temporarily influence gingival display.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult individuals with a gummy smile who provide consent for photographic documentation
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
value of gummy smile visibility using artificial intelligence algorithms | 1 month
  gummy smile visibility

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Turgut Çankaya, Phd DDS, Study Director — Gazi University
Locations (1):
- Zeynep Turgut Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: CSR
Time Frame: The data will become available whitin 1 month and will be available one year